CLINICAL TRIAL: NCT01157104
Title: A Phase I, Double-Blind, Multiple-Dose Study to Evaluate the Pharmacokinetic Drug-Drug Interaction Between IDX320 and IDX184 in Healthy Subjects
Brief Title: A Drug-Drug Interaction Study Evaluating the Combination of IDX320 and IDX184 in Healthy Participants (MK-6844-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 6844-002; IDX-07A-002 (Other: Idenix)
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Hepatitis C
Keywords: HCV; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — IDX320; IDX184

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- IDX320 + PBO → IDX320 + IDX184 (Experimental): 400 mg IDX320 and IDX184 matching placebo (PBO) once daily for 7 days; followed by 400 mg IDX320 and 100 mg IDX184 once daily for 7 days
  Interventions: Drug: IDX320; Drug: IDX184; Drug: IDX184 placebo
- IDX184 + PBO → IDX184 + IDX320 (Experimental): 100 mg IDX184 and IDX320 matching PBO for 7 days; followed by 100 mg IDX184 and 400 mg IDX320 for 7 days
  Interventions: Drug: IDX320; Drug: IDX184; Drug: IDX320 placebo
- IDX320 PBO + IDX184 PBO (Placebo Comparator): IDX320 matching PBO + IDX184 matching PBO for 14 days
  Interventions: Drug: IDX184 placebo; Drug: IDX320 placebo

INTERVENTIONS:
Drug: IDX320 — IDX320 400 mg in tablets (8x50 mg) administered orally once daily
  Arms: IDX184 + PBO → IDX184 + IDX320; IDX320 + PBO → IDX320 + IDX184
Drug: IDX184 — IDX184 100 mg in capsules (2x50 mg) administered orally once daily
  Arms: IDX184 + PBO → IDX184 + IDX320; IDX320 + PBO → IDX320 + IDX184
Drug: IDX184 placebo — IDX184 matching placebo in capsules administered orally once daily
  Arms: IDX320 + PBO → IDX320 + IDX184; IDX320 PBO + IDX184 PBO
Drug: IDX320 placebo — IDX320 matching placebo in tablets administered orally once daily
  Arms: IDX184 + PBO → IDX184 + IDX320; IDX320 PBO + IDX184 PBO

SUMMARY:
This study is designed to evaluate the potential for a pharmacokinetic (PK) drug-drug interaction between IDX320 and IDX184 and to assess the safety and tolerability when the two drugs are administered in combination in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study, participants must meet the following requirements:

1. Must be a healthy male or female between 19 and 65 years of age with body mass index (BMI) between 18 and 35 kg/m2.
2. Must be a non-smoker.
3. Must agree to use an acceptable double-barrier method of birth control.
4. Must provide written informed consent after the study has been fully explained.

Exclusion Criteria:

Participants are not eligible if they meet any of the following:

1. Pregnant or breastfeeding.
2. History of clinically significant diseases, as determined by the investigator.
3. Safety laboratory abnormalities at screening which are clinically significant.
4. Positive screening test for hepatitis B virus, hepatitis C virus or human immunodeficiency virus (HIV).
5. Use of chronic prescription medications within 3 months, acute prescription medications within 14 days, or systemic over-the-counter (OTC) medications within 7 days of the starting the study.
6. Current abuse of alcohol or illicit drugs, or history of alcohol or illicit drug abuse within the preceding two years.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Area under the curve at steady state (AUCss) of plasma IDX320 | Days 1-7 pre-dose; Day 7: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20 hrs postdose; Days 8-14 pre-dose; Day 14: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hrs postdose
AUCss of plasma IDX184 | Days 1-7 pre-dose; Day 7: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20 hrs postdose; Days 8-14 pre-dose; Day 14: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hrs postdose
AUCss of plasma 2'-methylguanosine (2'-MeG) | Days 1-7 pre-dose; Day 7: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20 hrs postdose; Days 8-14 pre-dose; Day 14: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hrs postdose
Maximum observed concentration (Cmax) of plasma IDX320 | Days 1-7 pre-dose; Day 7: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20 hrs postdose; Days 8-14 pre-dose; Day 14: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hrs postdose
Cmax of plasma IDX184 | Days 1-7 pre-dose; Day 7: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20 hrs postdose; Days 8-14 pre-dose; Day 14: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hrs postdose
Cmax of plasma 2'-MeG | Days 1-7 pre-dose; Day 7: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20 hrs postdose; Days 8-14 pre-dose; Day 14: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hrs postdose
Trough concentration (Ctrough) of plasma IDX320 | Days 1-7 pre-dose; Day 7: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20 hrs postdose; Days 8-14 pre-dose; Day 14: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hrs postdose
Ctrough of plasma IDX184 | Days 1-7 pre-dose; Day 7: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20 hrs postdose; Days 8-14 pre-dose; Day 14: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hrs postdose
Ctrough of plasma 2"-MeG | Days 1-7 pre-dose; Day 7: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20 hrs postdose; Days 8-14 pre-dose; Day 14: 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hrs postdose

SECONDARY OUTCOMES:
Number of participants with an adverse event (AE) | Up to Day 19
Number of participants who discontinued treatment due to an AE | Up to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC